CLINICAL TRIAL: NCT05213130
Title: The Relationship Between Blood Donation and Subjective Well-being
Brief Title: Blood Donation and Subjective Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, Senior Investigator, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Blood donation and well-being
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Blood Donation; Happiness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude-based intervention (Experimental): Participants in this group receive a standardized gratitude-based intervention immediately after completing whole-blood donation. The intervention consists of (1) a written gratitude reinforcement message acknowledging the donor's contribution and emphasizing the life-saving impact of their donation, and (2) a brief vignette illustrating how donated blood benefits patients in need. The purpose of this intervention is to enhance donors' subjective well-being and psychological need satisfaction by reinforcing their sense of autonomy, competence, and relatedness. Participants complete questionnaires at Time 1 (post-donation) and Time 2 (4-22 days later).
  Interventions: Other: Information
- No Message (No Intervention): Participants in this group complete the standard post-donation procedure and receive no additional message or vignette. They complete the same questionnaires at Time 1 (post-donation) and Time 2 (4-22 days later) as the Intervention group. This arm serves as the comparison condition for evaluating the effect of the gratitude-based intervention on subjective well-being and related psychosocial outcomes.

INTERVENTIONS:
Other: Information — A reminder to inform donors that their blood has saved patient's life in a questionnaire.
  Arms: Gratitude-based intervention

SUMMARY:
This study investigates the psychological effects of blood donation among adult donors at the Guangzhou Blood Center. The primary objective is to examine whether a brief gratitude-based intervention delivered after donation enhances donors' subjective well-being (SWB) and basic psychological need (BPN) satisfaction. Participants who complete a whole-blood donation are randomly assigned to either an Intervention group, receiving a standardized gratitude reinforcement message accompanied by a vignette emphasizing the life-saving impact of donation, or a Control group that receives no additional message. All participants complete questionnaires at Time 1 (immediately after donation) and at Time 2 (4-22 days later), assessing SWB and related psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed a whole-blood donation at the Guangzhou Blood Center during the study period.
* Able to read and understand the study materials and provide informed consent.
* Provided the correct answer to a control question in the questionnaire
* Provided their phone number.
* Donated blood was successfully supplied to the hospitals.

Exclusion Criteria:

* Whole blood donors with positive or suspicious serological results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 601 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Score of Subjective Well-Being at Time 2 | 4-22 days after donation
  Subjective well-being (SWB) is assessed at follow-up using a validated multi-item measure capturing life satisfaction and affective well-being.
  Affect-Adjective Scale (validated Chinese version): 9 items, each scored 1-7. Satisfaction with Life Scale (validated Chinese version): 5 items scored 1-7. An aggregate SWB score was calculated by standardizing and summing life satisfaction scores with positive affect scores and subtracting the negative affect score from them.
  Scores range from low to high levels of well-being. The primary objective is to evaluate whether exposure to the gratitude-based intervention leads to higher SWB relative to the control condition.

SECONDARY OUTCOMES:
Score of Subjective Well-being at Time 1 | Immediately after donation
  Baseline Subjective well-being (SWB) is measured using a validated multi-item measure capturing life satisfaction and affective well-being.
  Affect-Adjective Scale (validated Chinese version): 9 items, each scored 1-7. Satisfaction with Life Scale (validated Chinese version): 5 items scored 1-7. An aggregate SWB score was calculated by standardizing and summing life satisfaction scores with positive affect scores and subtracting the negative affect score from them.
  Scores range from low to high levels of well-being.
Score of Basic Psychological Needs Satisfaction at Time 1 | Immediately after donation
  Baseline basic psychological needs (BPN) satisfaction is measured using a 9-item Basic Psychological Needs Scale (validated Chinese version). The scale contains subscales for autonomy, competence, and relatedness, using a 7-point scale ranging from 1 (not at all true) to 7 (very much true). Each of the three subscales was averaged to form an index of general BPN satisfaction. This measure captures donors' immediate psychological experience following donation. Higher scores indicate greater psychological need satisfaction.
Score of Basic Psychological Needs Satisfaction at Time 2 | 4-22 days after donation
  The same basic psychological needs satisfaction (BPN) scale is administered at follow-up to examine changes after the intervention. It is measured using a 9-item Basic Psychological Needs Scale (validated Chinese version). The scale contains subscales for autonomy, competence, and relatedness, using a 7-point scale ranging from 1 (not at all true) to 7 (very much true). Each of the three subscales was averaged to form an index of general BPN satisfaction. Higher scores indicate greater psychological need satisfaction.
Score of Blood Donation Intention at Time 1 | Immediately after donation
  Intention to donate blood again in the future at Time 1 is measured using a single self-report intention item rated from 1 (very unlikely) to 7 (very likely), with higher scores indicating stronger intention to donate. The same item is administered at Time 1 and Time 2 to assess changes over time and to examine potential effects of the intervention on future donation motivation.
Score of Blood Donation Intention Score at Time 2 | 4-22 days after donation
  Intention to donate blood again in the future at Time 2 is measured using a single self-report intention item rated from 1 (very unlikely) to 7 (very likely), with higher scores indicating stronger intention to donate. The same item is administered at Time 1 and Time 2 to assess changes over time and to examine potential effects of the intervention on future donation motivation.
Re-Donation Rate within One Year | Up to 12 months after the initial donation
  Actual re-donation rate is obtained from the Guangzhou Blood Centre's donation records. The variable indicates whether the participant returned for another whole-blood or component donation within one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No